CLINICAL TRIAL: NCT02798575
Title: Detecting Chronic Obstructive Pulmonary Disease (COPD) Exacerbations and Need for Hospitalization With Software Analysis of Ventilators for Invasive Mechanical Ventilation
Brief Title: COPD Exacerbations
Status: Terminated | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-025
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: COPD
Keywords: COPD; invasive ventilation; exacerbation; home care; mechanical ventilation; unsuccessful weaning; ventilatory parameters
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples for arterial blood gas analyses
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Astral 150 ventilator — Patients indicative for invasive ventilation will receive the Astral 150 ventilator at the weaning station of the hospital. The ventilator will be set by the physician. Afterwards patients will be transferred into home care.

SUMMARY:
Detecting exacerbations to prevent a severe and / or to early treat an exacerbation is crucial in patients with COPD in order to prevent hospitalization. Patients with invasive mechanical ventilation outside the hospital have a high re-hospitalization rate which is associated with severe economic burden since those patients need to be treated mainly on an ICU or a respiratory ward being able to take care of invasive mechanical ventilation.

Recently, it has been shown that daily variations of parameters recorded by non-invasive ventilation (NIV) software are predictors of exacerbations in a cohort of COPD patients being treated outside the hospital with NIV [1]. These parameters were respiratory rate and percentage of respiratory cycles triggered by the patient.

The aim of the present study is to detect parameters recorded by the ventilator which are able to predict exacerbation and / or hospitalization in patients with COPD under invasive mechanical ventilation outside the hospital.

DETAILED DESCRIPTION:
The number of mechanically ventilated patients in the intensive care unit (ICU) is increasing due to a rise in the frequency of respiratory and cardiovascular diseases as well as demographical changes. As a result, there is a corresponding increase in the time required for the complex process of weaning from mechanical ventilation (MV). Weaning from MV contributes to up to 50% of the duration of respiratory support. Especially those patients with prolonged weaning (≥3 spontaneous breathing trials over ≥7 days) refer to a very complex patient group with either chronic co-morbidities (e.g. chronic obstructive pulmonary disease [COPD]) or extended treatment in the ICU as a result of acute conditions (e.g. septic or cardiogenic shock, acute respiratory failure) or other significant diseases.

Not all of these patients can be weaned from the ventilator. An increasing number of patients are in need for invasive mechanical ventilation following unsuccessful weaning. They often need special care regarding ventilatory support, management of tracheal secretion and muscular re-conditioning.

These patients, especially those with COPD, are at high risk for further exacerbations and have thus a high rate of re-hospitalization. An early detection of exacerbations to rapidly implement therapeutic interventions is a major goal in the management of patients with severe COPD but may need close contact to medical experts.

However, a physician-based structure for treating this specific patient group does not exist, so that these patients often have hospital treatment. This might be preventable if clinical determinants and ventilator parameters would be detected timely.

Home ventilators for invasive ventilation are provided with built-in software recording data such as respiratory rate (RR), percentage of respiratory cycles triggered by the patient (%Trigg), tidal volume and daily usage of the ventilator. A systematic assessment of variations in specific ventilator-based parameters may help to predict the risk of exacerbation in patients with COPD treated by home care.

In sum, the objective of this study is to assess whether day-to-day variation in these ventilatory parameters recorded by the ventilators can predict an imminent exacerbation or need for hospitalization in patients with COPD treated at home with invasive ventilation. This is supposed to be of major importance, both for the progression of the disease and for economic reasons regarding the health care system. The possibility of detecting exacerbations due to ventilator analysis might be a further step towards telemonitoring of ventilator-dependent patients

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with COPD indicative for invasive ventilation outside the hospital
2. Male or female aged > 18 years
3. Written informed consent prior to study participation by patient or legal representative

Exclusion Criteria:

1. Pregnant and lactating females
2. Indication for invasive ventilation outside the hospital due to other disease than COPD
3. Inability or Unwillingness to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD who are in need for invasive mechanical ventilation following unsuccessful weaning.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Occurence of an exacerbation of COPD | up to 12 months
  An exacerbation or unplanned hospitalization will be defined as following:
  Event 1: "Exacerbation without hospital admission" In case of administration of antibiotics and / or steroids by a general practitioner, this event will be defined as exacerbations of COPD.
  Event 2: "Critical exacerbation with hospital admission" In case of administration of antibiotics and / or steroids by a general practitioner and an additional hospitalization, this event will also be defined as a critical exacerbation.
  Event 3: "Hospital admission without exacerbation" In case of hospitalization for reasons other than exacerbation (e.g. patients dys-synchrony on ventilator, other somatic reasons), this event will also be defined and recorded.

SECONDARY OUTCOMES:
EXACT Pro Questionnaire | up to 12 months
  The questionnaire will be performed weekly by patients or legal representative in order to evaluate exacerbations and respiratory symptoms in clinical studies of COPD.
Arterial blood gas (ABG) | baseline, month 3, month 6 and month 12
  Blood samples for arterial blood gas analysis (ABG) will be performed at baseline, month 3, month 6 and month 12.
Evaluation of demographic data | baseline, month 3, month 6 and month 12
  Demographic data will be recorded and evaluated at baseline, follow up at month 3, month 6 and month 12.
Daily usage of ventilator (in hours) | up to 12 months
  Daily usage of ventilator will be recorded by the ventilator daily during home care. Analysis of the recorded data will be performed at month 3, month 6 and month 12.
Tidal volume | up to 12 months
  Tidal volume will be recorded by the ventilator daily during home care. Analysis of the recorded data will be performed at month 3, month 6 and month 12.
%Trigg cycled breaths | up to 12 months
  %Trigg cycled breaths will be recorded by the ventilator daily during home care. Analysis of the recorded data will be performed at month 3, month 6 and month 12.
Respiratory Rate (RR) | up to 12 months
  The RR will be recorded by the ventilator daily during home care. Analysis of the recorded data will be performed at month 3, month 6 and month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Bickenbach, Dr., Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Borel JC, Pelletier J, Taleux N, Briault A, Arnol N, Pison C, Tamisier R, Timsit JF, Pepin JL. Parameters recorded by software of non-invasive ventilators predict COPD exacerbation: a proof-of-concept study. Thorax. 2015 Mar;70(3):284-5. doi: 10.1136/thoraxjnl-2014-206569. Epub 2015 Jan 12. PMID 25582449
- [Background] Zilberberg MD, de Wit M, Pirone JR, Shorr AF. Growth in adult prolonged acute mechanical ventilation: implications for healthcare delivery. Crit Care Med. 2008 May;36(5):1451-5. doi: 10.1097/CCM.0b013e3181691a49. PMID 18434911
- [Background] Lilly CM, Zuckerman IH, Badawi O, Riker RR. Benchmark data from more than 240,000 adults that reflect the current practice of critical care in the United States. Chest. 2011 Nov;140(5):1232-1242. doi: 10.1378/chest.11-0718. Epub 2011 Aug 25. PMID 21868469
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Leidy NK, Wilcox TK, Jones PW, Murray L, Winnette R, Howard K, Petrillo J, Powers J, Sethi S; EXACT-PRO Study Group. Development of the EXAcerbations of Chronic Obstructive Pulmonary Disease Tool (EXACT): a patient-reported outcome (PRO) measure. Value Health. 2010 Dec;13(8):965-75. doi: 10.1111/j.1524-4733.2010.00772.x. PMID 20659270